CLINICAL TRIAL: NCT00207454
Title: Optimizing Strategies to Improve STD Partner Services
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: State University of New York - Downstate Medical Center (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: CDC-NCHSTP-3197; R30/CCR219136-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Chlamydia Trachomatis; Neisseria Gonorrhoeae
Keywords: Partner Referral; Social Cognitive Intervention; Partner Delivered Medication

INTERVENTIONS:
Behavioral: Social Cognitive Counseling

SUMMARY:
This research tests the effectiveness of a social cognitive intervention (with option of patient-delivered medication) geared toward increasing patient referral of partners.

DETAILED DESCRIPTION:
This is a four-year study involving longitudinal data collection for 800 men and women recruited from four clinics in Brooklyn, NY. Participants were eligible for enrollment at any of the study sites if diagnosed as having C trachomatis or N gonorrhoeae genital infection or if they have an STD syndrome likely to be related to either of these pathogens (i.e., males with NGU). Consenting patients were randomly assigned to receive either standard-of-care patient referral for partner notification (N = 350), a social-cognitive intervention geared toward increasing patient referral (N = 350), or the social-cognitive intervention with an option of patient-delivered medication (N = 100). Evaluation activities include an interviewer administered measure provided at baseline, one month, and six months, a screen for N gonorrhoeae and C trachomatis using urine-based ligase chain reaction screening (Abbott LCx) at baseline and six months, and medical chart abstraction at one and six months.

ELIGIBILITY:
Inclusion Criteria:

* Any individual presenting at study sites with STD-related symptoms who receives a microbiologic diagnosis with N gonorrhoeae and/or C trachomatis will be eligible for study participation if they meet the following criteria: 1) are 18 years of age or older; 2) have been sexually active in the previous two months; 3) are able to understand English or Spanish; 4) have resided within the catchment area for at least one year prior to enrollment; 5) plan to remain in the area through the course of the study period. .

Exclusion Criteria:

* Any potential participant deemed by a provider or member of the study staff to have psychological impairment, brought on by drug use or some other illness, to an extent that it would affect the ability to understand or provide informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800
Dates: Start 2001-06; Study Completion 2005-08

PRIMARY OUTCOMES:
Partner notification 1 month
Repeat Infection 6 month

SECONDARY OUTCOMES:
Intent to notify partner baseline post-test
Changes in relationship 1 month, 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Tracey Wilson, PhD, Principal Investigator — State University of New York - Downstate Medical Center
Locations (1):
- STD Clinic at Kings County Hospital Center (KCHC)., Brooklyn, New York, United States